CLINICAL TRIAL: NCT01140009
Title: A Randomized, Blinded, Placebo-controlled, Cross-over Study of the Safety and Immunogenicity of Trivalent, Inactivated Influenza Vaccine for 2010-2011
Brief Title: Safety and Protectiveness of the Seasonal Influenza Vaccine for 2010-2011
Acronym: PCIRNRT06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H10-01356
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: Vaccine; Seasonal Influenza vaccine; Influenza vaccine; Vaccine safety; Vaccine immunogenicity; Fluviral 2010/11
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Placebo Comparator): FLuviral 2010/11Tri-valent Seasonal Influenza Vaccine (TIV)1st; saline placebo 10 days later
  Interventions: Biological: Fluviral 2010/11 Tri-valent Seasonal Influenza vaccine
- Group 2 (Placebo Comparator): Saline placebo 1st; Fluviral 2010/11 Tri-valent Seasonal Influenza Vaccine (TIV)10 days later
  Interventions: Biological: Fluviral 2010/11 Tri-valent Seasonal Influenza vaccine

INTERVENTIONS:
Biological: Fluviral 2010/11 Tri-valent Seasonal Influenza vaccine — Vaccination of .05mL of Fluviral vaccine will be injected once at either visit 1 or 2 depending upon randomization in the deltoid muscle of the non-dominant arm
  Arms: Group 1
Biological: Fluviral 2010/11 Tri-valent Seasonal Influenza vaccine — Vaccination of .05mL of Fluviral vaccine will be injected once at either visit 1 or 2 depending upon randomization in the deltoid muscle of the non-dominant arm
  Arms: Group 2

SUMMARY:
The seasonal influenza vaccination program for 2010-2011 will be the first to follow the H1N1 pandemic of 2009. Many Canadians either had the H1N1 infection or the adjuvanted H1N1 vaccine. Both H1N1 infection and adjuvanted vaccine produced strong immune responses which could last for some time.

The seasonal influenza vaccine for this fall will be a "normal" product once again, without adjuvant. It will contain 3 strains of killed, split-apart viruses that might circulate this winter, including the H1N1 pandemic strain. It is theoretically possible that giving the H1N1-containing seasonal vaccine to people who still have some immunity to H1N1 virus could result in more frequent side-effects. However, there is no good evidence that pre-existing immunity to a strain in the vaccine does increase side-effects. In short, there could be nothing out of the ordinary this fall but it would be prudent to check this before public flu vaccination programs begin.

DETAILED DESCRIPTION:
This study will assess the safety of seasonal influenza vaccination in people who had the adjuvanted H1N1 vaccine last year. It will also measure residual immunity to the H1N1 virus and immune responses to the seasonal vaccine. It will be carried out before the new vaccine is released for general use so that we have an accurate picture of vaccine safety and responses for other Canadians.

A total of 320 adults (64 at each site) 20 to 59 years old, are being asked to participate in this study. A research nurse will conduct a telephone screening with potential participants to determine if they are eligible for the study. Volunteers must have had adjuvanted H1N1 vaccine before January 31, 2010.

The study involves 2 vaccination visits 10 days part. At one visit seasonal vaccine will be given and at the other a placebo vaccine will be given. Which vaccine is given first will be determined by random chance, the details of which will not be released until study end. After each vaccination, there will be contacts 1 and 7 days later for a description of any symptoms experienced. A blood sample will be requested at the first and last visits (visit 3) to measure immune responses to the seasonal vaccine.

The study will take 21-38 days to complete, depending upon the vaccination sequence and availability. Total time required to take part is about 2.5 hours. The 3 study visits will occur at a clinic in Vancouver, Calgary, Ottawa, Montreal or Quebec City.

Each subject will be asked to keep daily notes of any changes at the injection site (pain, redness, swelling) and any general symptoms (such as headache, tiredness, body aches), including your oral temperature, for 7 days after each vaccination. Major health changes will be assessed for 21 days post 'vaccination'

A special Safety Board will review the results of the first vaccinations and advise whether it is reasonable to continue the study or not.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Can and will comply with the requirements of the protocol
* Age 20-59 years at Visit 1
* Receipt of one dose of Arepanrix (adjuvanted H1N12009 vaccine, GSK) in 2009 documented by written record or attested by a confident personal recollection (window for vaccination will be 1 October 2009 to January 31, 2010).

Exclusion Criteria:

* Systemic hypersensitivity to hens' eggs or to any other Fluviral S/F vaccine component such as thimerosal
* History of a life-threatening reaction to any influenza vaccine
* Receipt of non-study TIV for the 2010-2011 season
* Receipt of any live vaccine within 4 weeks or inactivated vaccine within one week of study entry or planned administration of any non-study vaccines during the study period
* Thrombocytopenia or any bleeding disorder that contraindicates IM injection or blood collection
* Pregnancy, at any stage of gestation
* Receipt of blood or any blood-derived products within 3 months prior to Visit 1
* Chronic illness at a stage that could interfere with trial participation (stable health conditions are acceptable, such as diabetes, lung disease, heart conditions etc)
* History of Guillain-Barre syndrome
* Immune compromise as a result of illness or immunosuppressive medication
* Participation in any other research study involving a non-approved drug or medical device
* Any other condition that may interfere with ability to comply with trial procedures, including abuse of alcohol, drug addiction or imposed confinement
* Current febrile illness or oral temperature of ≥ 38.0 °C

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of 2010-2011 seasonal trivalent vaccine (TIV) | 12 weeks
  To evaluate the safety of 2010-2011 seasonal trivalent vaccine (TIV) in a convenience sample of adults being re-vaccinated with H1N12009 antigen, as soon as vaccine becomes available so as to inform subsequent use of the vaccine in public programs.
To measure immune responses to each component of TIV | 12 weeks
  To measure immune responses to each component of TIV prior to and following seasonal vaccination to assess the immunogenicity of the new TIV vaccine.
To observe the persistence of anti-HAI responses to H1N12009 | 12 weeks
  To observe the persistence of anti-HAI responses to H1N12009 in a subset of subjects previously studied after vaccination with adjuvanted pandemic vaccine in late 2009 and to compare their peak responses to H1N12009 after the pandemic and TIV vaccinations.

SECONDARY OUTCOMES:
Vaccine-attributable rates of the observed adverse events | 12 weeks
  The secondary safety outcomes will be the vaccine-attributable rates of the observed adverse events, both local and general,
Immunogenicity analysis performed on the according-to-protocol (ATP) cohort | 12 weeks
  The secondary immunogenicity outcome will be the immunogenicity analysis performed on the according-to-protocol (ATP) cohort, comprising subjects with complete data for the principal immunogenicity endpoints and no major protocol deviations. The key immunogenicity outcome will be whether the HAI antibody responses to each vaccine strain meet the EMEA/CHMP criteria (3) for seasonal TIV vaccine responses in adults <60 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, Dr., Principal Investigator — University of British Columbia; Simon Dobson, Dr., Study Director — University of British Columbia; Laura Sauve, Dr., Study Director — University of British Columbia; Tobias Kollmann, Dr., Study Director — University of British Columbia; Keswadee Lapphra, Dr., Study Director — University of British Columbia; Brian Ward, Dr., Study Director — McGill University Health Centre - Vaccine Study Centre; Marc Dionne, Dr., Study Director — Unité de Recherche en Santé Publique (CHUQ); Vladimir Gilca, Dr., Study Director — Unité de Recherche en Santé Publique (CHUQ); Gaston DeSerres, Dr., Study Director — Unité de Recherche en Santé Publique (CHUQ); Curtis Cooper, Dr., Study Director — The Ottawa Hospital Research Institute, University of Ottawa; Otto Vanderkooi, Dr., Study Director — ACHIEVE Research, Alberta Children's Hospital, University of Calgary and Alberta Health Services; James Kellner, Dr., Study Director — ACHIEVE Research, Alberta Children's Hospital, University of Calgary and Alberta Health Services; Judy MacDonald, Dr., Study Director — ACHIEVE Research, Alberta Children's Hospital, University of Calgary and Alberta Health Services
Locations (5):
- Canada (5):
  - ACHIEVE Research, Alberta Children's Hospital, Calgary, Alberta
  - Vaccine Evaluation Center, Vancouver, British Columbia
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - McGill University Health Centre - Vaccine Study Centre, Montreal, Quebec
  - Unité de Recherche en Santé Publique, Québec, Quebec

REFERENCES:
- [Derived] Skowronski DM, Janjua NZ, De Serres G, Purych D, Gilca V, Scheifele DW, Dionne M, Sabaiduc S, Gardy JL, Li G, Bastien N, Petric M, Boivin G, Li Y. Cross-reactive and vaccine-induced antibody to an emerging swine-origin variant of influenza A virus subtype H3N2 (H3N2v). J Infect Dis. 2012 Dec 15;206(12):1852-61. doi: 10.1093/infdis/jis500. Epub 2012 Aug 7. PMID 22872731